CLINICAL TRIAL: NCT06496334
Title: 3-D Computed Forensic Facial Reconstruction of Computed Tomography (CT) Scanned Skulls Using Human Facial Templates
Brief Title: Forensic Facial Reconstruction (FFR) From CT Scans
Status: Completed | Type: Observational
Sponsor: Queen Mary University of London (Other)
Collaborators: Ministry of Higher Education & Scientific Research (Egypt) (Unknown)
Responsible Party: Sponsor
Other Study IDs: Forensic Facial Reconstruction; Computed FFR using CT (Other: Queen Mary University of London)
Record Dates: First submitted 2014-07-11; First posted 2024-07-11 (Actual); Last update posted 2025-03-11 (Actual); Status verified 2025-03

CONDITIONS: Forensic Facial Reconstruction
Keywords: Forensic facial reconstruction

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Head CT scan: Adult Caucasian patients undergoing head CT scanning.

SUMMARY:
1. Reconstructing faces derived from CT scanned skulls using the average facial templates and employing computer facial reconstruction software programme.
2. Evaluating the accuracy of facial reconstructions by objective comparison between the reconstructed face and the CT scanned face.
3. Evaluating the accuracy of facial reconstructions by subjective assessment via 2 groups of individuals, experienced and inexperienced in facial images perception.

DETAILED DESCRIPTION:
1. Patients Recruitment Patients meeting the inclusion criteria are identified and recruited by the attending clinical staff at a private Diagnostic Radiology Center in Egypt after completing the relevant ethical and regulatory procedures.The study will include a minimum of 20 case studies.
2. Acquisition of CT Scanned Head Images CT images are acquired by a computed tomography scanner.
3. Segmentation (i.e extraction) of a 3D images of the skull from CT Digital Imaging and Communications in Medicine (DICOM) files: via 3D slicer software and Simpleware (CT segmenting software) trial software.
4. Selection of Average Face Templates For each studied case, the facial reconstruction will be conducted using an average Caucasian face template that matches the studied skull, in terms of sex and age group selected.
5. Facial Reconstruction is performed using the patient segmented skull image and its matching average face template, and employing the present computer software program.
6. Segmentation (i.e extraction) of a 3D images of the face surface from CT DICOM files.
7. Objective Assessment of Facial Reconstructions for each case via objective surface superimposition between the extracted 3D facial image and the 3D reconstructed face using Robin's surface viewer software.

   The sum of square differences (SSD) between the superimposed images will be calculated as an indication of the goodness of fit of the reconstructed face with the CT scanned face. The measured differences will then be correlated with the sum of scores given to each reconstructed face by subjective assessment.
8. Subjective Assessment by Volunteers Assessors Volunteer assessors will be approached in an attempt to evaluate the accuracy of the resulting reconstructed images. Two groups of assessors will be recruited; the first assessors will be experts with professional experience in face image identification (n=5), and the second group will comprise of participants inexperienced in forensic facial identification. The latter will be recruited from staff and students of Queen Mary University of London (QMUL) (n=20-30). All participants will be asked to sign a written confidentiality agreement.

   1. Face Pool Test Construction The aim of face pool test in the present study is to assess the ability of observers to identify a target subject from a face pool of similar subjects. The face pool will be formed of computer generated faces, in 5 views (frontal, right lateral and left lateral, right ¾ and left ¾), included the extracted CT face of the target and these faces will be compared to the target facial reconstruction. Each observer will be asked to select one image from the test faces that best matches the target reconstructed face.
   2. Resemblance Test Construction This test aims to compare and assess the similarity between the facial reconstruction and the CT face of a target subject using rating/ranking scale. Each observer will be asked to rate the target reconstructed face from 0 to 10 according to its resemblance to the target CT face , where 0 = no resemblance and 10 = highest resemblance. Facial reconstructions of all cases will be ranked by the total resemblance scores given by all observers to each reconstruction.
9. Statistical analysis of the results via spearman's Rank coefficient to assess and compare:

   1. Facial reconstructions ranks given by the 2 groups of observers to assess the influence of previous experience in face identification on the ability of the observer to assess the accuracy of forensic facial reconstructions.
   2. Facial reconstructions ranks given by subjective and objective assessment methods, thus compare the validity of both methods in assessing the accuracy of forensic facial reconstructions.

ELIGIBILITY:
Inclusion Criteria:

1. Caucasian ethnicity. Caucasian ethnicity is the general physical type of some or all of the populations of Europe, North Africa, the Horn of Africa, Western Asia, Central Asia and South Asia.
2. Above 16 years of age.
3. Able to understand and willing to sign the written Informed Consent Form.
4. Able and willing to follow the protocol requirements.
5. Undergoing CT scanning of the head for medical or clinical purposes.
6. A full CT head series is undertaken.

Exclusion Criteria:

1. Ethnic background other than Caucasian.
2. Less than 16 years old.
3. Unable to understand or refusing to sign the written Informed Consent.
4. Unable or refusing to follow the protocol requirements.
5. Unclear or incomplete head CT scan images.
6. Disfiguring bone or soft tissue deformity or scans with implantable devices (i.e. eye, head and neck, or cardiac).

Ages: 16 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: 1. This study will involve conducting facial reconstruction of 3-D human skull images acquired from head CT scanning of living patients in a private Diagnostic radiology center in Egypt.
  2. The resulting facial reconstructions will then be assessed by 2 groups of volunteer participants; experts and non-experts in the field of facial identification respectively.
Sampling Method: Non-Probability Sample
Enrollment: 2 (Actual)
Dates: Start 2014-05-28 (Actual); Primary Completion 2015-04-30 (Actual); Study Completion 2015-04-30 (Actual)

PRIMARY OUTCOMES:
The percentage of correct identifications and resemblance scores of the target reconstructed faces by human assessors. | 3 years

SECONDARY OUTCOMES:
The influence of previous experience in the field of facial image recognition and perception on the identification of the reconstructed faces. | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Dalia AS Abdou, MSc, Principal Investigator — PhD student, Queen Mary University of London; Peter Vanezis, MD, PhD, Principal Investigator — Professor of Forensic Medical Sciences, Queen Mary University of London; Atholl Johnston, PhD, Principal Investigator — Professor of Clinical Pharmacology, Queen Mary University of London
Locations (1):
- Barts School of Medicine and Dentistry, Queen Mary University of London, London, United Kingdom